CLINICAL TRIAL: NCT01711918
Title: Domperidone for the Treatment of Chronic Nausea and Vomiting Secondary to Gastroparesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ron Schey (Other)
Responsible Party: Sponsor-Investigator, Ron Schey, Clinical Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Domperidone
Record Dates: First submitted 2012-10-18; First posted 2012-10-22 (Estimated); Results first posted 2016-12-19 (Estimated); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Patients With Gastroparesis Who Have Failed Standard Therapy
Keywords: gastroparesis; domperidone; nausea; vomiting
MeSH Terms: conditions — Gastroparesis; Nausea; Vomiting | interventions — Domperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Domperidone (Experimental): Participants will received domperidone at a dose of 10mg given up to three times per day
  Interventions: Drug: Domperidone

INTERVENTIONS:
Drug: Domperidone — oral tablet; dose is 10mg per tablet given up to 3 times daily.

SUMMARY:
To provide oral domperidone to patients between the ages of 18 and 60 years of age, according to the investigator's judgment, a prokinetic effect is needed for the relief of severe gastroparesis. We have defined severe gastroparesis as 1) positive gastric emptying scintigraphy (more than 10% residue at 4 hours), 2) nausea, 3) early satiety, 4) abdominal pain. We will recruit patients for two years and the patients will be given domperidone for up to two years.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female
2. Age 18 - 60
3. Symptoms or manifestation secondary to gastroparesis such as vomiting, nausea, the feeling you are full after you start eating, and abdominal pain.
4. Subjects must have a comprehensive evaluation to eliminate other causes of their symptoms which includes gastric emptying scintigraphy, esophagogastroduodenoscopy (EGD), and the patient's subjective symptoms.
5. Subject has signed informed consent for the administration of domperidone that informs the patient of potential adverse events
6. Female subjects must be:

   1. surgically sterile (have had a hysterectomy or bilateral oophorectomy, or tubal ligation)
   2. if sexual active, practicing an effective method of birth control such as hormonal prescription oral contraceptives, progesterone implants or injections, contraceptive patch, intrauterine device, or maintenance of a monogamous relationship with a male partner who has been surgically sterilized by vasectomy. A double barrier method such as condoms, diaphragms, or cervical caps with spermicidal foam, cream, or gel may be used as a method of birth control

Exclusion Criteria:

1. History of, or current, arrhythmias including ventricular tachycardia, ventricular fibrillation, atrial fibrilation and Torsade des Pointes, subjects with minor forms of ectopy (PACs) are not necessarily excluded
2. Clinically significant bradycardia, sinus node dysfunction, or heart block. Prolonged QTc (QTC>450 milliseconds for males, QTc>470 milliseconds for females)
3. Clinically significant electrolyte disorders
4. Gastrointestinal hemmorrhage or obstruction
5. Presence of a prolactinoma (prolactin-releasing pituitary tumor)
6. Pregnant or breast feeding female
7. Known allergy to domperidone The following medications are prohibited during the study: antidepressants: doxepin, clomipramine, amopxapine, trazodone, venlafaxine, nefazodone, fluvoxamine, paroxetine, fluoxetine, sertraline, amitriptyline, maprotiline, desipramine, nortriptyline, trimipramine, imipramine, protriptyline; anti-psychotics: haloperidol, chlorpromazine, chlorpromazine pimozide, sertindole, quetiapine, mesoridazine, perphenazine, lfluphenazine, promazine, trifluoperazine; anti-emetics: prochlorperazine, thioridazine, promethazine, mesoridazine, theiethylperazine, perphazine, dolasetron, dronabinol, droperidol; anti-infective agents: erythromycin, clarithromycin, troleandomycin, norfloxcin, quinine sulfate, quinupristin and dalfopristin, pentamidine, sparfloxacin, grepafloxacin, azithromycin, ofloxacin, levofloxacin; anti-fungal agents: fluconazole, itraconazole, ketoconazole, miconazole, terconazole, ticonazole, butaconazole; antivirals: foscarnet; protease inhibitors: indinavir, amprenavir, ritonavir, nelfinavir, squinavir; antihypertensives: nicardipine, isradipine, moexipril/HCTZ; calcium channel blockers: verapamil, diltiazem, deltiazem/enalapril, verapamil/trandolapril, tocainide, bepridil; anti-arrhythmics: disopyramide, quinidine, procainamide, flecainide, sotalol, bretylium, amiodarone, ibutilide, moricizine; diueretics: bumetanide, furosemide, torsemide, etharcrynic acid, chlorothiazide, indapamide; antilipemics: probucol, bepridil, mibefradil; hematological agents: cilostazol; respiratory agents: zafirlukast, salmetrol; gastrointestinal agents: cimetidine, cisapride; antidiarrheal: octreotide; antihistamines: azelastine, clemastine; migraine treatment: naratriptan, sumatriptan, zolmitriptan; antimalarial: halofantrine; muscle relaxants: tizanidine; narcotic dependence: levomethadyl; miscellaneous: tamoxifen, warfarin, phenytoin, ziprasidone, risperidone, formoterol fumarate, sildenafil; drugs that prolong the QT Interval: albuterol, alfuzosin, amantadine, amisulpride, amphetamine, arsenic trioxide, astemizole, atazanavir, atomoxetine, chloral hydrate, chloroquine, ciprofloxacin, citalopram, clozapine, cocaine, dexmethylphenidate, diphenhydramine, dobutamine, dofetilide, dopamine, dronedarone, ephedrine, epinephrine, eribulin, escitalopram, famotidine, felbamate, fenfluramine, fingolimod, fosphenytoin, galantamine, gatifloxacin, gemifloxacin, granisetron, iloperidone, isoproterenol, lapatinib, levalbuterol, lisdexamfetamine, lithium, metaproterenol, methadone, methylphenidate, midodrine, moxifloxacin, nilotinib, norepinephrine, ondansetron, oxytocin, paliperidone, perflutren lipid microspheres, phentermine, phenylephrine, phenylpropanolamine, protriptyline, pseudoephedrine, ranolazine, ritodrine, toxithromycin, sibutramine, solifenacin, sunitinib, tacrolimus, telithromycin, terbutaline, terfenadine, tolterodine, trimethoprim-sulfa, vandetanib, vardenafil, voriconazole.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2012-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Domperidone
Started | 9
Completed | 7
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Domperidone
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Improvement of Overall Symptoms Based on Likert Scale
Description: A subject will be considered a responder, if they report on a 6 point Likert scale that when compared to baseline, their symptoms are either 'somewhat better or markedly better'.
Time Frame: Baseline and End of study (2 years or last visit if patient withdraws)
Measure: Count of Participants; unit: Participants
Arm/Group | Domperidone
Number analyzed (Participants) | 7
Participants | 2

2. Secondary Outcome: Improvement of Nausea Based on Likert Scale
Description: as for outcome 1
Time Frame: Baseline and End of study (2 years or last visit if patient withdraws)
Measure: Count of Participants; unit: Participants
Arm/Group | Domperidone
Number analyzed (Participants) | 7
Participants | 2

3. Secondary Outcome: Improvement of Vomiting Based on Likert Scale
Description: as for outcome 1
Time Frame: Baseline and End of study (2 years or last visit if patient withdraws)
Measure: Count of Participants; unit: Participants
Arm/Group | Domperidone
Number analyzed (Participants) | 7
Participants | 2

4. Secondary Outcome: Improvement of Abdominal Bloating or Distention Based on Likert Scale
Description: as for outcome 1
Time Frame: Baseline and End of study (2 years or last visit if patient withdraws)
Measure: Count of Participants; unit: Participants
Arm/Group | Domperidone
Number analyzed (Participants) | 7
Participants | 2

5. Secondary Outcome: Improvement of Premature Abdominal Fullness After Meals Based on Likert Scale
Description: as for outcome 1
Time Frame: Baseline and End of study (2 years or last visit if patient withdraws)
Measure: Count of Participants; unit: Participants
Arm/Group | Domperidone
Number analyzed (Participants) | 7
Participants | 1

ADVERSE EVENTS:
Arm/Group | Domperidone
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 5/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Domperidone (N=7)
Allergic Reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Partial Bowel Obstruction (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Heartburn (Gastrointestinal disorders) | 1 (1)
Hypophosphatemia (Blood and lymphatic system disorders) | 1 (1)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Ruptured Right Ovarian Cyst (Reproductive system and breast disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Ear and labyrinth disorders) | 1 (1)
Shaking (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Hand Tingling (Nervous system disorders) | 1 (1)
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dry Mouth (General disorders) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chest Palpitations (Cardiac disorders) | 1 (1)
Elevated ALT (Hepatobiliary disorders) | 1 (1)
Elevated AST (Hepatobiliary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes